CLINICAL TRIAL: NCT02236052
Title: Immunogenicity, Safety and Tolerability of a Plant-Derived Seasonal Virus-Like Particles (VLP) Quadrivalent Influenza Vaccine in the Elderly Population
Brief Title: Immunogenicity, Safety and Tolerability of a Plant-Derived Seasonal VLP Quadrivalent Influenza Vaccine in the Elderly Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicago (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CP-Q13VLP-008
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections
Keywords: Influenza; Human; RNA Virus Infections; Immunologic; Immunogenic Factors; Physiological Effects of Drugs; Virus diseases; Orthomyxoviridae Infections; Infection
MeSH Terms: conditions — Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections; Influenza, Human; Orthomyxoviridae Infections; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Non-adjuvanted low dose of quadrivalent VLP vaccine (Experimental): A single non-adjuvanted low dose of quadrivalent VLP vaccine
  Interventions: Biological: Non-adjuvanted low dose of quadrivalent VLP vaccine
- Non-adjuvanted medium dose of quadrivalent VLP vaccine (Experimental): A single non-adjuvanted medium dose of quadrivalent VLP vaccine
  Interventions: Biological: Non-adjuvanted medium dose of quadrivalent VLP vaccine
- Non-adjuvanted high dose of quadrivalent VLP vaccine (Experimental): A single non-adjuvanted high dose of quadrivalent VLP vaccine
  Interventions: Biological: Non-adjuvanted high dose of quadrivalent VLP vaccine
- Adjuvanted low dose of quadrivalent VLP vaccine (Experimental): A single low dose of quadrivalent VLP vaccine mixed with Alhydrogel®
  Interventions: Biological: Adjuvanted low dose of quadrivalent VLP vaccine
- Adjuvanted high dose of quadrivalent VLP vaccine (Experimental): A single high dose of quadrivalent VLP vaccine mixed with Alhydrogel®
  Interventions: Biological: Adjuvanted high dose of quadrivalent VLP vaccine
- Placebo (Placebo Comparator): A single dose of Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Non-adjuvanted low dose of quadrivalent VLP vaccine — A single non-adjuvanted low dose of quadrivalent VLP vaccine
  Arms: Non-adjuvanted low dose of quadrivalent VLP vaccine
Biological: Non-adjuvanted medium dose of quadrivalent VLP vaccine — A single non-adjuvanted medium dose of quadrivalent VLP vaccine
  Arms: Non-adjuvanted medium dose of quadrivalent VLP vaccine
Biological: Non-adjuvanted high dose of quadrivalent VLP vaccine — A single non-adjuvanted high dose of quadrivalent VLP vaccine
  Arms: Non-adjuvanted high dose of quadrivalent VLP vaccine
Biological: Adjuvanted low dose of quadrivalent VLP vaccine — A single low dose of quadrivalent VLP vaccine mixed with Alhydrogel®
  Arms: Adjuvanted low dose of quadrivalent VLP vaccine
Biological: Adjuvanted high dose of quadrivalent VLP vaccine — A single high dose of quadrivalent VLP vaccine mixed with Alhydrogel®
  Arms: Adjuvanted high dose of quadrivalent VLP vaccine
Biological: Placebo — A single dose of placebo
  Arms: Placebo

SUMMARY:
This is a multiple sites phase II trial, randomized, observer-blind, dose ranging, placebo-controlled study to evaluate the immunogenicity, safety, and tolerability of a single intramuscular injection of plant-based Seasonal VLP Quadrivalent Influenza Vaccine administered in elderly subjects (50 years old and more).

A total of four hundred fifty (450) subjects will be randomized in six (6) groups of 75 subjects to receive one injection of either a non-adjuvanted low, medium or high dose level of VLP, a low or high dose level of VLP of the quadrivalent VLP influenza vaccine combined with Alhydrogel® as adjuvant or the placebo preparation (100 millimolar (mM) phosphate buffer + 150 mM sodium chloride (NaCl) + 0.01% Tween 80)

DETAILED DESCRIPTION:
This study will use cohort staggering (slow enrollment) for 3 non-adjuvanted dose levels (low, medium, high dose level of VLP per strain), 2 adjuvanted dose levels (low or high dose level of VLP per strain) and a placebo-controlled group divided in 3 cohorts:

* Cohort 1: Approximately one hundred and thirty-eight (138) subjects will be randomized and dosed as follows: seventy-five (75) subjects with the lowest non-adjuvanted dose of the quadrivalent VLP vaccine, nineteen (19) subjects with the medium non-adjuvanted dose of the quadrivalent VLP vaccine, nineteen (19) subjects with the lowest adjuvanted dose of the quadrivalent VLP vaccine and twenty-five (25) subjects with a placebo. The 7-day safety data after the immunization will be collected by the clinical staff and will be reviewed by the Data and Safety Monitoring Board (DSMB). The DSMB consisting of the PIs, the Sponsor's Medical Officer and 3 external medical advisors (voting members); the members will determine if the clinical sites are allowed to continue with the immunization of the second cohort.
* Cohort 2: Approximately one hundred and seventy-five (175) subjects will be randomized and dosed as follows: fifty-six (56) subjects with the medium non-adjuvanted dose quadrivalent VLP vaccine, fifty-six (56) subjects with the lowest adjuvanted dose quadrivalent VLP vaccine, nineteen (19) subjects with the highest adjuvanted dose quadrivalent VLP vaccine, nineteen (19) subjects with the highest non-adjuvanted dose quadrivalent VLP vaccine and twenty-five (25) subjects with a placebo. The 7-day safety data after the immunization will be collected by the clinical staff and reviewed by the DSMB prior to allowing immunization of the third cohort.
* Cohort 3: Approximately one hundred and thirty-seven (137) subjects will be randomized and dosed as follows: fifty-six (56) subjects with the highest adjuvanted dose, fifty-six (56) subjects with the highest non-adjuvanted dose and twenty-five (25) subjects with a placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, 50 years of age or older.
2. BMI of ≥18 and ≤32.
3. Give his/her consent to participate in this study (by signing the informed consent form). In the opinion of the Investigator, competence and willingness to provide written, informed consent for participation after reading the informed consent form. The subject must have adequate opportunity to discuss the study with an Investigator or qualified designee.
4. Healthy as judged by the Investigator or designee and determined by general physical examination, vital signs, clinical laboratory tests, and medical history conducted no more than 90 days prior to study vaccine administration. Subjects with a pre-existing chronic disease will be allowed to participate if the disease is stable and, according to the Investigator's judgment, the condition is unlikely confound the results of the study or pose additional risk to the subject by participating in the study. Stable disease is defined as no new onset of exacerbation of pre-existing chronic disease 6 months prior to immunization. Based on Investigator's judgment, a subject with more recent stabilisation of a disease may still be eligible.
5. Comprehension of the study requirements, expressed availability for the required study period, ability to attend scheduled visits, accessible by phone on a consistent basis.
6. If female, have a negative serum pregnancy test result at screening and negative urine pregnancy test on Day 0 prior to immunization.
7. Female of childbearing potential must use an effective method of contraception for 1 month prior to immunization and agrees to continue employing adequate birth control measures for at least 60 days post-immunization. Moreover, she must have no plan to become pregnant for at least 2 months post-immunization. Abstinent subjects should be asked what method(s) they would use, should their circumstances change, and subjects without a well-defined plan should be excluded.

   The following relationship or methods of contraception are considered to be effective:
   * Hormonal contraceptives (e.g., injectable, topical [patch], estrogenic vaginal ring, etc.);
   * Intra-uterine device (IUD) with or without hormonal release;
   * Male partner using a condom plus spermicide or sterilized partner (at least 1 year prior to immunization);
   * History of credible abstinence (self-reported);
   * Heterosexual abstinence at least 60 days post-immunization;
   * Female partner.
8. Non-childbearing females defines as:

   * Surgically-sterile (defined as bilateral tubal ligation or hysterectomy performed more than 1 month prior to immunization);
   * Post-menopausal (absence of menses for 24 consecutive months and age consistent with natural cessation of ovulation).

Exclusion Criteria:

1. According to Investigator's opinion, presence of significant acute or chronic, uncontrolled medical or neuropsychiatric illness. "Uncontrolled" is defined as:

   1. Requiring a new medical or surgical treatment within one month prior to study vaccine administration which would interfere with vaccine evaluation or study completion (subject requiring medical or surgical treatment that would not interfere with evaluation [e.g., minor knee surgery, cataracts, etc.] would be eligible);
   2. Requiring a change in medication dosage in one month prior to study vaccine administration due to uncontrolled symptoms or drug toxicity (elective dosage adjustments in stable subjects are acceptable).
2. Any medical or neuropsychiatric condition or any history of excessive alcohol use or drug abuse which, in the Investigator's opinion, would render the subject unable to provide informed consent or unable to provide valid safety observations and reporting.
3. Any autoimmune disease or any confirmed or suspected immunosuppressive condition or immunodeficiency including history of human immunodeficiency virus (HIV) infection, Hepatitis B or C, or the presence of lymphoproliferative disease.
4. Administration of any vaccine (including any other influenza vaccine) within 30 days prior to study enrolment or planned administration within the period from the vaccination up to blood sampling at Day 21 or within 30 days prior to blood sampling at Day 201. Immunization on an emergency basis will be evaluated in a case-by-case by the Investigator.
5. Administration of any adjuvanted or investigational influenza vaccine within 1 year prior to study enrolment or planned administration prior to the end of this trial (Day 201). Administration of any 'standard', not adjuvanted influenza vaccine (e.g., live attenuated Trivalent Inactivated Influenza Vaccine (TIV) or Quadrivalent Inactivated Vaccine (QIV) vaccine IN or split TIV or QIV vaccine by either intra-dermal or intramuscular route) prior to the 30-day exclusion period mentioned above would be acceptable.
6. Use of any investigational or non-registered product within 30 days prior to study enrolment or planned use during the study period. Subjects may not participate in any other investigational or marketed drug study while participating in this study (approximately 7-12 months [depending when subjects undergo screening session and Day 201 visit]).
7. Treatment with systemic glucocorticoids at a dose exceeding 10 mg of prednisone per day, or equivalent for more than 7 consecutive days or for 10 or more days in total, within one month of study vaccine administration, any other cytotoxic or immunosuppressant drug, or any immunoglobulin preparation within 3 months of vaccination. Routine use of standard doses of nasal or inhaled glucocorticoids is allowed.
8. Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving prophylactic anti-platelet medications, e.g., low-dose aspirin (no more than 325 mg/day), and without a clinically apparent bleeding tendency are eligible. Subjects treated with new generation drugs that will not increase risk of intramuscular bleeding (such as clopidogrel) are also eligible.
9. History of allergy to any of the constituents of the VLP quadrivalent study vaccine, Alhydrogel® (aluminum hydroxide) or to the phosphate buffered saline (PBS; used as placebo), or tobacco allergy.
10. History of anaphylaxis reaction to any food, medication or bee sting.
11. Any history of severe asthma (e.g., status asthmatic, hospitalization for asthma control) or recurrent asthma episodes requiring medical attention in the last 3 years (≥ 1 episode/year).
12. Continuous use of anti-histamines in the last 4 weeks prior to immunization or use of anti-histamines 48 hours prior to study immunization.
13. Have a rash, dermatological condition, tattoos, muscle mass, or any other abnormalities at injection site which may interfere with injection site reaction rating.
14. Have received a blood transfusion within 90 days prior to study vaccination.
15. If female, have a positive or doubtful pregnancy test prior to immunization or lactating females.
16. Vital sign abnormalities (systolic blood pressure and/or diastolic blood pressure, heart rate). Although a vital signs measurement is out of the acceptable ranges, a subject may be included in the study based on Investigator's judgment. Presence of any febrile illness (including oral temperature (OT) ≥38.0˚C within 24 hours prior to immunization). Such subjects may be re-evaluated for enrolment after resolution of illness.
17. Cancer or treatment for cancer within 3 years of study vaccine administration. Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible. Persons with treated and uncomplicated basal cell carcinoma of the skin are eligible. Person with non-treated, non-disseminated local prostate cancer are eligible.
18. Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2014-07-16 (Actual); Primary Completion 2015-06-17 (Actual); Study Completion 2015-06-17 (Actual)

PRIMARY OUTCOMES:
Immunogenicity | 21 days after injection
  Immunogenicity will be assessed by Geometric mean titers (GMTs) of Hemagglutination Inhibition (HI) antibodies against the vaccine strains on Days 0 and 21 and assessed by measuring geometric mean fold rise, seroconversion rate and seroprotection rate. Follow-up serology samples for GMTs will be collected at Day 201.
Solicited systemic and local reactions | 21 days after injection
  Safety and tolerability will be assessed by the rate, severity and relationship to vaccination of solicited and unsolicited adverse events post-vaccination. A 6-month follow-up period will be performed.

SECONDARY OUTCOMES:
Immunogenicity (against vaccine strains and heterologous strains) | 21 days after injection
  Immunogenicity will be evaluated by Geometric mean titers (GMTs) of microneutralization (MN) antibodies (Days 0 and 21) against the vaccine strains and assessed by measuring Geometric mean fold rise ans seroconversion rate. Cross-reactivity of antibodies induced by a single dose of the quadrivalent VLP vaccine will also be assessed and measured by HI and microneutralization (MN) antibody titers for heterologous influenza strains. This will be assessed using the measure of Geometric mean fold rise, seroconversion rate and seroprotection rate (for HI only).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Libman, MD, Principal Investigator — MUHC-Vaccine Study Centre; Guy Boivin, MD, Principal Investigator — Centre de recherche-CHU de Québec; Richard Larouche, MD, Principal Investigator — inVentiv Health Clinique
Locations (3):
- Canada (3):
  - MUHC-Vaccine Study Centre, Pierrefonds, Quebec
  - Centre de recherche-CHU de Québec, Québec
  - inVentiv Health Clinique, Québec

REFERENCES:
- [Result] Pillet S, Couillard J, Trepanier S, Poulin JF, Yassine-Diab B, Guy B, Ward BJ, Landry N. Immunogenicity and safety of a quadrivalent plant-derived virus like particle influenza vaccine candidate-Two randomized Phase II clinical trials in 18 to 49 and >/=50 years old adults. PLoS One. 2019 Jun 5;14(6):e0216533. doi: 10.1371/journal.pone.0216533. eCollection 2019. PMID 31166987